CLINICAL TRIAL: NCT01696006
Title: Perfusion CT Registry
Acronym: Perfusion CT
Status: Completed | Type: Observational
Sponsor: Young-Hak Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Young-Hak Kim, MD, PhD, Young-Hak Kim, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV 2012-04
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: perfusion computed tomography; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether coronary perfusion computed tomography is effective in the treatment of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 20
* Patient who has a coronary perfusion computed tomography

Exclusion Criteria:

* Unwillingness or inability to give informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General hospital
Sampling Method: Non-Probability Sample
Enrollment: 1059 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of coronary perfusion computed tomography | 5year
  Positive predictive value Negative predictive value Sensitivity Specificity

SECONDARY OUTCOMES:
Relationship between coronary perfusion computed tomography and fraction flow reserve | 5year
Relationship between coronary perfusion computed tomography and SPECT(nuclear imaging) | 5year
occurrence of the event after coronary perfusion computed tomography | 5year
  Death Myocardial infarction coronary angiography Revascularization

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Asan Medical Center, Seoul, Songpa-Gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang university hospital, Bucheon-si
  - Dong-A university hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - ChonBuk National University Hospital, Jeonju
  - Inje university Pusan Paik hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Kwon O, Hwang HJ, Koo HJ, Yang DH, Kang HJ, Kim JA, Moon DH, Kim HS, Kang JW, Kim YH. Ischemic burden assessment of myocardial perfusion CT, compared with SPECT using semi-quantitative and quantitative approaches. Int J Cardiol. 2019 Mar 1;278:287-294. doi: 10.1016/j.ijcard.2018.12.046. Epub 2018 Dec 17. PMID 30587418
- [Derived] Kang SJ, Kweon J, Yang DH, Lee JG, Jung J, Kim N, Mintz GS, Kang JW, Lim TH, Park SW, Kim YH. Mathematically Derived Criteria for Detecting Functionally Significant Stenoses Using Coronary Computed Tomographic Angiography-Based Myocardial Segmentation and Intravascular Ultrasound-Measured Minimal Lumen Area. Am J Cardiol. 2016 Jul 15;118(2):170-6. doi: 10.1016/j.amjcard.2016.04.049. Epub 2016 May 5. PMID 27236253
- [Derived] Kang SJ, Yang DH, Kweon J, Kim YH, Lee JG, Jung J, Kim N, Mintz GS, Kang JW, Lim TH, Park SW. Better Diagnosis of Functionally Significant Intermediate Sized Narrowings Using Intravascular Ultrasound-Minimal Lumen Area and Coronary Computed Tomographic Angiography-Based Myocardial Segmentation. Am J Cardiol. 2016 Apr 15;117(8):1282-8. doi: 10.1016/j.amjcard.2016.01.022. Epub 2016 Jan 28. PMID 26892449